CLINICAL TRIAL: NCT05829083
Title: Asymmetric (DUET) Versus Conventional Nasal High Flow Interface for Management of Hypercapnic Patients With Mild to Moderate Acute Exacerbation of COPD: A Randomized, Crossover Clinical Trial
Brief Title: DUET Versus Standard Interface for Hypercapnic COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: Sotiria General Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Pantazopoulos, Assistant Professor of Emergency Medicine, Larissa University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 51886
Record Dates: First submitted 2023-03-09; First posted 2023-04-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: COPD Exacerbation; Hypercapnia; COPD
MeSH Terms: conditions — Hypercapnia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypercapnic COPD patient - Asymmetric or conventional nasal high flow cannula (Experimental): Patients with acute exacerbation of COPD and mild to moderate hypercapnic respiratory failure will be randomized to NHF oxygen therapy with asymmetric cannula OR conventional cannula
  Interventions: Device: Asymmetric nasal cannula - DUET; Device: Conventional nasal high flow cannula
- Hypercapnic COPD patient - Conventional or asymmetric nasal high flow cannula (Active Comparator): Patients with acute exacerbation of COPD and mild to moderate hypercapnic respiratory failure will be randomized to NHF oxygen therapy with conventional cannula or Asymmetric cannula
  Interventions: Device: Asymmetric nasal cannula - DUET; Device: Conventional nasal high flow cannula

INTERVENTIONS:
Device: Asymmetric nasal cannula - DUET — DUET asymmetric nasal high flow interface that fits best to the patients' nostrils (size: one nostril of the patient should be fully occluded)
  Patients will be crossed-over between the 2 interventions
Device: Conventional nasal high flow cannula — Well-established conventional nasal high flow cannula (size: medium)
  Patients will be crossed-over between the 2 interventions

SUMMARY:
The goal of this clinical trial is to compare the new asymmetric nasal high flow interface with the conventional high flow nasal cannula in patients with COPD exacerbation.

The main questions the study aims to answer are:

• Does the use of the asymmetric interface lead to:

1. A greater decrease in the patients' carbon dioxide
2. A greater decrease in respiratory rate and less dyspnea
3. Less need for advanced oxygen therapy measures
4. Same tolerance and comfort
5. Lower heart rate and blood pressure

Participants will be asked to:

Wear the asymmetric and conventional cannulas for 3 hours each with a 30 minute gap in-between. Arterial blood samples and various clinical parameters will be collected throughout the study period.

Researchers will compare the effect of asymmetric versus conventional cannulas to answer the aforementioned questions.

DETAILED DESCRIPTION:
Methods Study design and setting A randomized crossover clinical trial will be conducted at the University General Hospital of Larissa and Sotiria Thoracic Diseases Hospital of Athens. The order of therapy will be allocated using sequentially numbered, sealed envelopes not prepared by the study staff. It is not possible for the researchers or the patients to be blinded, due to the research design. Patients presenting to the emergency medicine department of the aforementioned hospitals with acute exacerbation of COPD will be screened for suitability. Consent to participate in the trial will be obtained from the patient or next of kin and the study will be conducted according to ICH-GCP and clinical trial regulations. The results of the study will be presented based on the CONSORT 2010 statement for randomized crossover trials.

Hypothesis The investigators hypothesize that patients on DUET asymmetric nasal high flow interface will generate higher external PEEP and will achieve a better clearance of CO2 compared to conventional NHF interface, leading to less inspiratory effort, less work of breathing and thus in reduction of pCO2 levels.

Study population and interventions Patients considered eligible for the study will be those (1) presenting to the emergency department with (2) acute exacerbation of COPD (defined as any worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to change in medication) with (3) mild-to-moderate acute hypercapnic respiratory failure (defined as 7.35>pH>7.25 and arterial CO2 tension (PaCO2) >45 mmHg).

Patients will be excluded if they meet one or more of the following criteria: acute on chronic hypercapnic respiratory failure, severe facial deformity, facial burns, fixed upper airway obstruction and any of the following criteria for imminent intubation and invasive mechanical ventilation (i.e. respiratory or cardiac arrest, diminished consciousness (Glasgow coma score <8), psychomotor agitation inadequately controlled by sedation, massive aspiration, persistent inability to remove respiratory secretions, severe haemodynamic instability unresponsive to fluids and vasoactive drugs, severe ventricular or supraventricular arrhythmias and life threatening hypoxaemia).

Fifty patients with acute exacerbation of COPD and mild to moderate hypercapnic respiratory failure will receive NHF oxygen therapy. Twenty-five patients will be randomly assigned to first receive NHF oxygen therapy with the largest DUET asymmetric NHF interface that fits best to the patients' nostrils, followed by medium size conventional NHF interface. Twenty-five patients will be randomly assigned to receive NHF oxygen therapy with medium size conventional NHF interface first, followed by the largest DUET asymmetric NHF interface that fits best to the patients' nostrils. During the study period, all patients will be studied in a semi-recumbent position and monitoring equipment will be applied. All patients will receive NHF therapy with the initial setting of flow at 60 lt/min, temperature at 37°C and FiO2 adjusted to maintain SpO2 between 88-92%. The NHF device and consumables will be the same for all patients (AIRVO 3, Fisher & Paykel Healthcare Ltd., Auckland, New Zealand).

Patients will receive the first randomized therapy for 3 hours (NHF therapy with DUET or conventional NHF interface), followed by a 30 min washout period of conventional oxygen therapy to control for the carry-over effect, after which they will cross over to the second therapy for 3 hours (NHF therapy with the largest DUET or conventional medium size NHF interface).

At any study point, if patient discomfort and/or deterioration or lack of improvement of the abovementioned physiologic variables occur, the researcher-attending physician will be free to switch the patient to NIV or invasive mechanical ventilation.

Data collection A case report form will be filled for each study participant. Demographic data including sex, age, weight, height, most recent pulmonary function testing and any concomitant health problems will be documented. Arterial blood gases (ABGs), vital signs (systolic and diastolic arterial pressure, heart rate), respiratory variables (respiratory rate, accessory muscle use, thoracoabdominal asynchrony), dyspnea score (with the Borg scale) and any pulmonary or extrapulmonary complications will be assessed. Researchers will also record patient's comfort by assessing the following: machine noise levels, mouth dryness and general perception of tolerance using a visual analogue scale from 0 (no inconvenience due to noise, no dryness, no discomfort) to 10 (maximum inconvenience due to noise, maximum dryness, maximum discomfort).

Pulse oximetry and calibrated transcutaneous CO2 monitoring will be attached and monitored continuously during the study period. A bio-impedance surface sensor will be placed and calibrated to measure noninvasively and continuously respiratory rate, tidal volume and minute ventilation (ExSpiron 2Xi, Respiratory motion, Inc., Waltham,MA).

The abovementioned measurements including ABGs will be collected at baseline, at the end of first randomized therapy, at the end of the washout period and at the end of the second therapy.

The cut-off values of the examined physiologic parameters indicating poor outcome with NHF are SpO2<88% not corrected with supplemental oxygen, respiratory rate >35 breaths·min-1, thoraco-abdominal asynchrony and auxiliary respiratory muscle use, worsening of hypercapnia and acidaemia, indicating further respiratory muscle fatigue and sequential organ failure assessment score >4.

ELIGIBILITY:
Inclusion Criteria:

* acute exacerbation of COPD (defined as any worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to change in medication)
* mild-to-moderate acute hypercapnic respiratory failure (defined as 7.35>pH>7.25 and arterial CO2 tension (PaCO2) >45 mmHg)

Exclusion Criteria:

* acute on chronic hypercapnic respiratory failure
* severe facial deformity, facial burns, fixed upper airway obstruction
* indication for imminent intubation and invasive mechanical ventilation (i.e. respiratory or cardiac arrest, diminished consciousness (Glasgow coma score <8)
* psychomotor agitation inadequately controlled by sedation
* massive aspiration
* persistent inability to remove respiratory secretions
* severe haemodynamic instability unresponsive to fluids and vasoactive drugs
* severe ventricular or supraventricular arrhythmias
* life threatening hypoxaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Arterial PCO2 | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Change in PCO2

SECONDARY OUTCOMES:
Respiratory rate | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Change in respiratory rate
Invasive or non-invasive mechanical ventilation | At the end of hospitalization (assessed up to 6 months), researchers will note if the patient needed invasive or non-invasive mechanical ventilation
  Need for Invasive or non-invasive mechanical ventilation
Tolerance | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Subjective tolerance of patients using visual analog scale (Score range: 0-10, higher scores indicate higher levels of tolerance)
Comfort | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Subjective comfort of patients using visual analog scale (Score range: 0-10, higher scores indicate higher levels of comfort)
Heart rate | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Patients' heart rate
Blood pressure | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Patients' blood pressure
Dyspnea | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Subjective dyspnea levels
Tidal volume | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Measurement of the amount of air that enters the lung per breath
Minute ventilation | Immediately before and after the application of 3 hours of nasal high flow therapy (3 hours for each cannula type)
  Measurement of the amount of air that enters the lungs per minute

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gourgoulianis, Ph.D., Study Chair — Larissa University Hospital
Locations (2):
- Greece (2):
  - Sotiria General Hospital, Athens
  - University Hospital of Larissa, Larissa

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 1 year of study completion
Access Criteria: Reasonable request

REFERENCES:
- [Background] Ischaki E, Pantazopoulos I, Zakynthinos S. Nasal high flow therapy: a novel treatment rather than a more expensive oxygen device. Eur Respir Rev. 2017 Aug 9;26(145):170028. doi: 10.1183/16000617.0028-2017. Print 2017 Sep 30. PMID 28794144
- [Background] Pantazopoulos I, Daniil Z, Moylan M, Gourgoulianis K, Chalkias A, Zakynthinos S, Ischaki E. Nasal High Flow Use in COPD Patients with Hypercapnic Respiratory Failure: Treatment Algorithm & Review of the Literature. COPD. 2020 Feb;17(1):101-111. doi: 10.1080/15412555.2020.1715361. Epub 2020 Jan 22. PMID 31965868
- [Background] Papalampidou A, Bibaki E, Boutlas S, Pantazopoulos I, Athanasiou N, Moylan M, Vlachakos V, Grigoropoulos V, Eleftheriou K, Daniil Z, Gourgoulianis K, Kalomenidis I, Zakynthinos S, Ischaki E. Nasal high-flow oxygen versus noninvasive ventilation in acute exacerbation of COPD: protocol for a randomised noninferiority clinical trial. ERJ Open Res. 2020 Oct 19;6(4):00114-2020. doi: 10.1183/23120541.00114-2020. eCollection 2020 Oct. PMID 33123554
- [Background] Crimi C, Noto A, Madotto F, Ippolito M, Nolasco S, Campisi R, De Vuono S, Fiorentino G, Pantazopoulos I, Chalkias A, Libra A, Mattei A, Scala R, Clini EM, Ergan B, Lujan M, Winck JC, Giarratano A, Carlucci A, Gregoretti C, Groff P, Cortegiani A; COVID-HIGH Investigators. High-flow nasal oxygen versus conventional oxygen therapy in patients with COVID-19 pneumonia and mild hypoxaemia: a randomised controlled trial. Thorax. 2023 Apr;78(4):354-361. doi: 10.1136/thoraxjnl-2022-218806. Epub 2022 May 17. PMID 35580898